CLINICAL TRIAL: NCT03952390
Title: Study on the Effect of Renin-Angiotensin System on Thrombocytopenia in Patient With Sepsis
Brief Title: Effect of Renin-Angiotensin System on Platelet in Patient With Sepsis
Acronym: ERASPPWS
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XHEC-C-2017-080
Record Dates: First submitted 2019-01-15; First posted 2019-05-16 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2018-12

CONDITIONS: Sepsis
Keywords: thrombocytopenia,Renin-Angiotensin System,platelet
MeSH Terms: conditions — Sepsis; Thrombocytopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma seperated from venous blood via centrifugation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: healthy volunteers
  Interventions: Other: control
- sepsis: patients with sepsis
  Interventions: Other: sepsis

INTERVENTIONS:
Other: control
  Other Names: healthy volunteers
  Groups: control
Other: sepsis
  Other Names: patients with sepsis
  Groups: sepsis

SUMMARY:
As a common and serious medical condition , sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection , which is a major and familiar cause of death in intensive care units(ICU). As a frequent laboratory abnormality in patients with sepsis , thrombocytopenia on intensive care unit admission is independently associated with increased mortality in patients. Furthermore, a low platelet count is a marker with further significance , which is always used for evaluating the prognosis of patients. Herein, this study aimed to investigate the effect of renin-angiotensin system on thrombocytopenia in patient with sepsis and explore the possible underlying molecular mechanisms.

DETAILED DESCRIPTION:
Sepsis should be defined as life-threatening organ dysfunction caused by a dysregulated host response to infection. According to the Centers for Disease Control and Prevention, sepsis occurs in 1.5 million Americans annually and it causes more than 250,000 deaths annually in the United States alone. Thrombocytopenia is a frequent laboratory abnormality in patients with sepsis. Sequential [Sepsis-related] Organ Failure Assessment (SOFA) score of 2 points or more represents organ dysfunction . As the index of coagulation , platelet count is involved in SOFA . The changes of quality and quantity in platelet is closely associated with the morbidity and mortality of infectious diseases . Furthermore , thrombocytopenia is independently related with increased mortality in severe sepsis patients . Therefore , rectify of thrombocytopenia is of significant role to prevent potentially life-threatening complications in patients with sepsis. Currently , donor-derived platelet transfusion is the only treatment of severe thrombocytopenia seen in sepsis . However , platelets used in the clinic is associated with lots of concerns , for example , sufficient availability , quality , and complications due to immunologic and/or infectious issues . So , it is necessary and urgent to focus our efforts on the development of therapeutic agents to overcome our dependence on donor-derived platelets for transfusion .

Deriving from megakaryocytes , platelets are anucleate , having only cytoplasmic components imparted by megakaryocytes residing in the bone marrow,circulating in the bloodstream and having an important role in the body because of their functions in hemostasis , thrombosis , inflammation , and vascular biology . There are numerous reasons why thrombocytopenia often accompany patients with sepsis , such as platelet-vessel wall interaction , excessive consumption of platelet in DIC and platelet activation . Furthermore, research indicates that the intrinsic machinery for programmed cell death (apoptosis) regulates the life span of the anucleate platelet. Besides, several mechanisms have been proposed to explain the platelet apoptosis ,among which reactive oxygen sepsis(ROS) appears to play critical role.

More studies have shown that the renin-angiotensin-aldosterone system(RAAS) is activated in sepsis,providing an important physiologic mechanism to preserve volume status and vascular tone. As the main effect factor of the RAAS, angiotensin II plays a key role in several biological processes, including apoptosis,coagulation ,cell growth, and inflammatory response in addition to its classical hemodynamic function of regulating arterial blood pressure.Numerous researches claimed , angiotensin II (Ang II) has been associated with organ failures and mortality by promoting the generation of a large amount of intracellular ROS. However, no studies have shown the relation between Ang II-related ROS and thrombocytopenia during sepsis.

Therefore, the investigators hypothesized that Ang II , by promoting the generation of a large amount of intracellular ROS , plays a critical role in the development of thrombocytopenia during sepsis.In the present study, the investigators will analyze the mechanism of platelet apoptosis during sepsis, and explore whether angiotensin II receptor blockers could protect ROS induced platelet apoptosis, which is helpful for prevention and treatment of thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection.

  • Organ dysfunction can be identified as an acute change in total SOFA score ≥2 points consequent to the infection.
* The baseline SOFA score can be assumed to be zero in patients not known to have preexisting organ dysfunction.
* ASOFA score ≥2 reflects an overall mortality risk of approximately 10% in a general hospital population with suspected infection. Even patients presenting with modest dysfunction can deteriorate further,emphasizing the seriousness of this condition and the need for prompt and appropriate intervention, if not already being instituted.

  * In lay terms, sepsis is a life-threatening condition that arises when the body's response to an infection injures its own tissues and organs.
  * Patients with suspected infection who are likely to have a prolonged ICU stay or to die in the hospital can be promptly identified at the bedside with qSOFA, ie, alteration in mental status, systolic blood pressure ≥100 mm Hg, or respiratory rate ≥22/min.
  * Septic shock is a subset of sepsis in which underlying circulatory and cellular/metabolic abnormalities are profound enough to substantially increase mortality.
  * Patients with septic shock can be identified with a clinical construct of sepsis with persisting hypotension requiring vasopressors to maintain MAP ≥65 mm Hg and having a serum lactate level >2 mmol/L (18mg/dL) despite adequate volume resuscitation. With these criteria,hospital mortality is in excess of 40%.

Abbreviations: MAP, mean arterial pressure; qSOFA, quick SOFA; SOFA: Sequential[Sepsis-related] Organ Failure Assessment.

Exclusion Criteria:

* Pregnant or lactation period.
* Age <18 years or >85 years.
* Receiving chemotherapy, steroid or immunosuppressive agents recently.
* Receiving any drugs that affect Renin-Angiotensin-System(RAS),sunch as Angiotensin Converting Enzyme Inhibitor(ACEI),Angiotensin Receptor Blockers(ARB)，diuretics，calcium channel blockers and other antihypertensives within two weeks .
* Receiving oral contraceptives within twelve weeks.
* Enrollment before resuscitation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with sepsis
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Platelet Count of Blood Sample | 20-60min
  The platelet count of venous blood samples collected from patients with sepsis was measured by Blood routine instrument,Beckman CoulterLH750.
The Plasma Renin Activity of Blood Sample | 20-60min
  Venous blood samples were collected in ethylenediaminetetraacetic acid (EDTA),dimercaptopropanol and 8 - hydroxyquinoline sulfate plus blood collection tubes, followed by centrifugation to separate plasma from venous blood samples.The plasma renin activity of venous blood samples collected from patients with sepsis was measured by Iodine[125I]AngiotensinⅡRadioimmunoassay Kit.
The Plasma Concentration of AngiotensinⅡ in Blood Sample | 20-60min
  Venous blood samples were collected in ethylenediaminetetraacetic acid (EDTA) ,dimercaptopropanol and 8 - hydroxyquinoline sulfate plus blood collection tubes, followed by centrifugation to separate plasma from venous blood samples.The plasma concentration of angiotensinⅡ in venous blood samples collected from patients with sepsis was measured by Iodine[125I]AngiotensinⅡRadioimmunoassay Kit.

SECONDARY OUTCOMES:
Correlation Coefficient (r) Between Platelet Count and The Plasma Renin Activity | 20-60min
  GraphPad Prism5 software were used to analysis the correlation coefficient (r) between platelet count and the plasma renin activity.If p value is less than 0.05, then its change is statically significant.
Correlation Coefficient (r) Between Platelet Count and The Plasma Concentration of AngiotensinⅡ | 20-60min
  GraphPad Prism5 software were used to analysis the correlation coefficient (r) between platelet count and the plasma concentration of angiotensinⅡ.If p value is less than 0.05, then its change is statically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Lai Jiang, chief doctor, Study Chair — Xinhua Hospital affiliated to Medicine school,Shanghai Jiaotong University
Locations (1):
- Department of Anesthesia, Shanghai Xinhua hospital, Shanghai, Shanghai Municipality, China